CLINICAL TRIAL: NCT04957329
Title: Department of Ophthalmology, Rigshospitalet-Glostrup Valdemar Hansens Vej 13, 2600 Glostrup, Denmark
Brief Title: Effect of Benzalkonium Chloride Preserved and Preservative-free Latanoprost Eye Drops on Conjunctival Goblet Cells
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Laboratoires Thea (Industry)
Responsible Party: Principal Investigator, Anne Hedengran Nagstrup, Department of ophthalmology, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WP3; 2019-001642-18 (EudraCT Number)
Record Dates: First submitted 2021-06-22; First posted 2021-07-12 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Intervention Model Description: each subject will be treated with a BAK-preserved eye drop in one eye and PF-eye drops in the other eye for 3 months.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAK-preserved (Active Comparator): Xalatan eye drop
  Interventions: Drug: Xalatan
- Preservative-free (Active Comparator): Monoprost eye drop
  Interventions: Drug: Monoprost

INTERVENTIONS:
Drug: Xalatan — Eye drop
  Other Names: BAK-preserved latanoprost
  Arms: BAK-preserved
Drug: Monoprost — Eye drop
  Other Names: Preservative-free latanoprost
  Arms: Preservative-free

SUMMARY:
a randomized, investigator-blind, interventinal study will compare the effect of benzalkonium-chloride (BAK) preserved and preservative-free (PF) eye drops on conjunctival goblet cells.

DETAILED DESCRIPTION:
The investigators will conduct a randomized, investigator-blind, interventinal study on 28 subjects. Each subject will apply a benzalkonium-chloride (BAK) preserved eye drop (Xalatan) in one eye and a preservative-free (PF) eye drop (Monoprost) in the other for 3 months. Which eye gets which treatment is randomized. Before and after treatment a conjunctival print will be made and the effect of the eye drops on goblet cell density will be evaluated along with effect on the intraocular pressure.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18years
2. Danish speaking
3. Open angle glaucoma or ocular hypertension
4. Average intraocular pressure equal to or above 22 mmHg

Exclusion Criteria:

a. history of significant eye diseae (including okular trauma) other than open angle glaucoma and ocular hypertension d. treatment with steroids within the last 3 months from inclusion e. Significant untreated systemic disease such as hypertension, heart failure, diabetes mellitus, stroke, lung disease and autoimmune diseases. Diseases are not reason for exclusion if they are well treated or does not need treatment g. pregnant or breast feeding h. women using unsafe anticonception i. allergy towards trial medication j. patients who cannot cooperate in eye examination k. ocular surface defects l. need for polytherapy in glaucoma treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Goblet cell density | 3 months
  Change in goblet cell density

SECONDARY OUTCOMES:
Intraocular pressure | 3 months
  change in intraocular pressure
Ocular surface | 3 months
  change in oxford scheme grading
Mucin content in tear film | 3 months
  change in mucin concentration
Cytokines in tear film | 3 months
  change in concentration of detectable interleukins e.g. interleukin 6
Ocular surface disease index evaluation | 3 months
  Change in OSDI

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Kolko, MD, PhD, Principal Investigator — Department of ophthalmology, rigshospitalet-Glostrup
Locations (2):
- Denmark (2):
  - Department of ophthalmology, rigshospitalet.glostrup, Glostrup Municipality, Danmark
  - Department of drug design and pharmacology, University of Copenhagen, Copenhagen

IPD SHARING:
Plan to Share IPD: No